CLINICAL TRIAL: NCT00005875
Title: Phase II Evaluation of RFS 2000 (9-Nitro-Camptothecin, 9NC) in Metastatic Melanoma
Brief Title: Nitrocamptothecin in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067911; SUPERGEN-RFS2000-10; MDA-DM-98237
Record Dates: First submitted 2000-06-02; First posted 2004-04-13 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-09

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and toxicity of nitrocamptothecin in patients with metastatic melanoma.

OUTLINE: Patients are stratified according to disease (choroidal vs nonchoroidal). Patients receive oral nitrocamptothecin daily on days 1-5. Treatment continues weekly for at least 8 weeks (2 courses) in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 28-74 patients (14-37 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic melanoma Choroidal (no prior chemotherapy required) OR Nonchoroidal No more than 3 chemotherapy regimens Bidimensionally measurable disease No symptomatic uncontrolled CNS involvement including extensive brain metastases, spinal cord compression, or meningeal carcinomatosis Not eligible for treatment protocol of higher priority

PATIENT CHARACTERISTICS: Age: Over 16 Performance status: Zubrod 0-2 Life expectancy: Greater than 8 weeks Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Transaminase no greater than 3 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 1 year after study No serious concurrent illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Show-Li Sun, MD, Study Chair — Astex Pharmaceuticals, Inc.
Locations (1):
- SuperGen, Incorporated, Dublin, California, United States